CLINICAL TRIAL: NCT00952016
Title: A Non-randomised Phase II Trial of Methotrexate in Metastatic Colorectal Cancer With MSH2 Deficiency
Brief Title: Methotrexate in Metastatic Colorectal Cancer With MSH2 Deficiency
Acronym: MESH
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recruitment - only 2 patients recruited.
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CCR3107
Record Dates: First submitted 2009-07-31; First posted 2009-08-04 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2009-08

CONDITIONS: Advanced Colorectal Cancer
Keywords: colorectal cancer; MSH2; metastatic
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Methotrexate — study subjects will receive methotrexate intravenously on day 1 and day 8 of a 3 weekly cycle.

SUMMARY:
To assess the efficacy of methotrexate in a genetically selected population of patients with advanced colorectal cancer, who have loss of a particular gene, MSH2. The efficacy of methotrexate will be evaluated by the proportion of cases that have a significant response to treatment (objective response rate).

DETAILED DESCRIPTION:
The study will involve treating 29 subjects with methotrexate given intravenously. All subjects will receive treatment; there is no control arm or randomisation. The subjects will be known to have deficiency of MSH2, or a mutation (genetic change) in MSH2 that stops it functioning normally. This can either be demonstrated by testing for loss of MSH2 protein in the tumour itself, or by the demonstration of a mutation in the MSH2 gene in the subject's blood.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of metastatic or locally recurrent colorectal carcinoma
* Aged 18 years or older
* Paraffin embedded histological material available for analysis
* Either confirmed loss of expression of MSH2 on immunohistochemistry IHC or confirmed mutation in MSH2 on gene sequencing
* Life expectancy of > 3 months

Exclusion Criteria:

* Previous treatment with methotrexate, either for malignant or non-malignant disease, except when methotrexate was given at low dose with other drugs to modify their effects
* Concomitant uncontrolled medical conditions
* Concomitant metastatic malignancy apart from non-melanotic skin cancers and carcinoma in situ of the uterine cervix in the last 10 years
* Any contraindication to treatment with methotrexate (as this will affect safety)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2009-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Objective response rate, to include complete response and partial response, as defined radiologically using RECIST (Response, Evaluation Criteria in Solid Tumours) on imaging CT scans performed during treatment.

SECONDARY OUTCOMES:
Disease stabilisation rate; progression free survival; 1 year survival and median overall survival; Quality of Life assessment; toxicity assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom